CLINICAL TRIAL: NCT03510676
Title: Innovative siroLimus seLf Expanding drUg-eluting Stent for the treatMent of perIpheral Disease: Evaluation of Safety aNd efficAcy. The ILLUMINA Study. (ILLUMINA)
Brief Title: The ILLUMINA Study. (ILLUMINA)
Acronym: ILLUMINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CID - Carbostent & Implantable Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P41302
Record Dates: First submitted 2018-04-04; First posted 2018-04-27 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NiTiDES (Experimental): Single arm
  Interventions: Device: NiTiDES

INTERVENTIONS:
Device: NiTiDES

SUMMARY:
The aim of the prospective, multicentre, single-arm study is to assess safety and efficacy of a drug eluting stent in Nitinol alloy (NiTiDES) in term of vessel patency and composite event-free survival rate up to two years follow-up in focal/medium length lesions in patients with ischemic obstruction of superficial femoral arteries or/and proximal popliteal arteries.

ELIGIBILITY:
Inclusion Criteria:

Clinical

* Patient must be over 18 years inclusive at the time of consent prior to participation in the study and must understand the purpose of this study and be willing to adhere to the study procedures described in this protocol;
* A female of childbearing potential may be enrolled, provided she has a negative pregnancy test at screening;
* Patient has signed and dated the informed consent;
* Patient has symptoms of peripheral arterial disease classified as Rutherford Category (2-4); patients with Rutherford Category 2 can be included only if a conservative and/or medication therapy was unsuccessful.
* Patient has a resting ABI <0.9 or at exercise if resting ABI is normal; patient with incompressible arteries (ABI >1.2) at rest or at exercise must have a toe-brachial index (TBI) <0.8.

Angiographic

* Patient has one documented stenotic or occluded atherosclerotic lesion (lesion length ≤ 14 cm) of the above-the-knee femoropopliteal artery, in one limb, that meet all of the inclusion criteria and none of the exclusion criteria;
* Patient has a de novo or restenotic lesion with >50% stenosis documented angiographically and no prior stent in the target lesion;
* The target lesion must be appropriately covered (margin of 5.0 mm on both sides of the stent) by one or two study stents (NiTiDES). Any occurred dissection of the target vessel must be treated with an additional stent (NiTiDES);
* Tandem lesions are allowed if the distance between 2 lesions is ≤ 3 cm and the total length of all lesions ≤ 14 cm;
* Guidewire successfully passed the lesion through the lumen.

Exclusion Criteria:

Clinical

* Patient is pregnant or breast-feeding;
* Patient is simultaneously participating in another investigational drug or device study;
* Patient has any planned surgical or interventional procedure within 30 days after the study procedure;
* Clinical conditions, disorders or allergies that limit the use of anti-platelet and/or anticoagulant therapy;
* Severe allergy to the contrast medium or drugs used during the procedure;
* Patients with known hypersensitivity or allergies to Sirolimus, fatty acids (such as stearic acid, palmitic acid, behenic acid) or the metal components of the stent (such as Nickel, Titanium and Tantalum);
* Serum creatinine > 2.5 mg/dl;
* Myocardial infarction within the 90 days prior to enrollment;
* Hypercoagulable state;
* Uncontrollable hypertension;
* Life expectancy < 12 months;
* Aneurysmal disease of abdominal aorta, iliac artery and popliteal artery;
* Gastrointestinal bleeding;
* Stroke within the 180 days prior to enrollment;
* Concomitant therapies such as: atherectomy, cryoplasty, scoring / cutting balloons.

Angiographic

* Patient has significant stenosis or occlusion of inflow tract not successfully treated before this procedure;
* Patient has had previous stenting of target vessel;
* Patient lacks at least one patent vessel of runoff with <50% stenosis throughout its course;
* Patient has untreated angiographically-evident thrombus in the target lesion;
* Patients intended to be treated with more than two stents in the target lesion unless additional stent required in case of dissection;
* Patient intended to receive different stent from NiTiDES in target lesion;
* Technically unsuccessful Percutaneous Transluminal Angioplasty (PTA) procedure, for example due to the impossibility of accessing the stenotic site with a delivery system
* Lesions considered untreatable with PTA or other interventional techniques;
* Inflow lesion ≥15 cm long or occlusion (any length) in the ipsilateral Iliac artery;
* Not successfully treated < 15 cm long inflow lesion in the ipsilateral iliac artery [Treatment of inflow lesion must precede patient enrollment and target lesion treatment. No Drug Eluting Stents (DES) and / or Drug Eluting Balloon (DEB) allowed for the treatment of inflow lesions];
* Lesions in contralateral Superficial Femoral Artery (SFA) that require intervention during the index procedure, or within 30 days after the index procedure. Lesions in contralateral SFA can be treated either >30 days prior to or > 30 days after the index procedure;
* Patient with stenosis adjacent to an aneurysmal lesion of diameter at least twice the lumen of the native vessel;
* Lesions localized in the two distal thirds of the popliteal artery (or at the knee joint, generally considered).

Others.

• Patients under judicial protection, tutorship or curatorship (for France only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Event-free survival rate from Major Adverse Events | 12 months after procedure
  Freedom from Clinical Events Committee (CEC) adjudicated Major Adverse Event (death, target limb amputation, target limb ischemia requiring surgical intervention or surgical repair of target vessel or clinically-driven target lesion revascularization) or worsening of the Rutherford score by 2 classes, or to class 5 or 6.
Primary patency (absence of clinically-driven target lesion revascularization or binary restenosis) | 12 months after procedure
  Primary patency is defined as absence of clinically-driven target lesion revascularization or binary restenosis; binary restenosis is defined as a peak systolic velocity ratio (PSVR) >2.4 (duplex evaluation)

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, Principal Investigator — Universitätsklinikum Leipzig, Germany
Locations (10):
- France (3):
  - Polyclinique Les Fleurs, Ollioules
  - Centre Privé Claude Galien, Quincy-sous-Sénart
  - Clinique Pasteur, Toulouse
- Germany (4):
  - Universitäts-Herzzentrum Freiburg, Bad Krozingen
  - St. Gertrauden Krankenhaus GmbH, Berlin
  - Universitätsklinikum Leipzig, Leipzig
  - Regiomed GefäBzentrum Sonneberg, Sonneberg
- Italy (3):
  - Maria Cecilia Hospital, Cotignola, Ravenna
  - San Raffaele Hospital, Milan
  - IRCCS Policlinico San Matteo, Pavia

REFERENCES:
- [Derived] Steiner S, Honton B, Langhoff R, Chiesa R, Kahlberg A, Thieme M, Zeller T, Garot P, Commeau P, Cremonesi A, Marone EM, Sauguet A, Scheinert D. 2-Year Results With a Sirolimus-Eluting Self-Expanding Stent for Femoropopliteal Lesions: The First-in-Human ILLUMINA Study. JACC Cardiovasc Interv. 2022 Mar 28;15(6):618-626. doi: 10.1016/j.jcin.2021.12.034. Epub 2022 Feb 23. PMID 35219622